CLINICAL TRIAL: NCT02919371
Title: Phase I/II Combined Alternating Sunitinib and Bevacizumab (Avastin®) in Advanced Renal Cell Carcinoma (CASA)
Brief Title: Combined Alternating Sunitinib and Bevacizumab (Avastin®) in Advanced Renal Cell Carcinoma (CASA)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Faisal Specialist Hospital & Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2141-102
Record Dates: First submitted 2015-03-24; First posted 2016-09-29 (Estimated); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sunitinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sunitinib and Bevacizumab Arm (Experimental): Phase I/II Combined Alternating Sunitinib and Bevacizumab (Avastin®) in Advanced Renal Cell carcinoma (CASA)Combined Alternating Sunitinib and Bevacizumab
  Interventions: Drug: Sunitinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Sunitinib — Oral therapy ( Anti-vascular endothelial growth factor Tyrosin Kinase Inhibitor): given as 50 mg daily from day 1 to day 28- cycle repeated every 42 days
  Other Names: Sutent
Drug: Bevacizumab — Monoclonal antibody against vascular endothelial growth factor: given intravenously on day 29 of each sunitinib cycle
  Other Names: Avastin

SUMMARY:
Combined sunitinib and bevacizumab in advanced renal cell carcinoma.

DETAILED DESCRIPTION:
This is a phase I/II trial of combined sunitinib and bevacizumab in advanced renal cell carcinoma ( CASBA) where Bevacizumab will be used only on day 29 of each 6 weeks sunitinib cycle.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed renal cell carcinoma with clear cell histology ( mixed histology with clear cell component is accepted)
2. Patient should have either locally advanced or metastatic disease
3. No prior anti-cancer therapy
4. Age ≥ 18 years
5. Life expectancy of 3 months or more
6. Measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) criteria version 1.1
7. Performance status 0-2 by ECOG scale
8. Patients with controlled brain metastasis are accepted
9. Adequate renal function: serum creatinine ≤ 2 times the institutional upper limit of normal
10. Adequate hepatic function: total bilirubin within normal institutional limits, serum AST and ALT levels ≤2 times the institutional upper limit of normal or ≤ 5 times the institutional upper limit of normal of elevated because of liver involvement
11. Coagulation (PT ≤ 1.5 times the institutional upper limit of normal)
12. Adequate hematological values: leukocyte count ≥3.0 x 109/L, an absolute neutrophil count ≥1.5 x 109/L, a platelet count ≥100 x 109/L and hemoglobin ≥ 9.0 g/dL
13. Urine dipstick for proteinuria <1+, patients discovered to have ≥ 1+ on dipstick urinanalysis at baseline should have urine protein/urine creatinine ratio ≤1
14. Singed written informed consent before enrolment
15. Patient should have unresectable disease ( for both the primary tumor and the metastasis)

Exclusion Criteria:

1. Inability to comply with the protocol therapy
2. Uncontrolled hypertension defined as BP more than 160 systolic and or more than 100 diastolic despite adequate treatment at the time of treatment initiation.
3. Severe cardiovascular disease (congestive heart failure NYHA III or IV, unstable angina pectoris, myocardial infarction, significant arrhythmias or Transient ischemic attack (TIA) or cerebrovascular accident (CVA) in the last 6 months
4. Major bleeding disorder, significant traumatic injury or recent major surgery within 28 days of starting therapy. Or minor surgery (FNA/Core biopsy) within 7 days of starting therapy
5. History of abdominal abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months
6. Pre-existing thyroid abnormality
7. Concurrent proarrhythmic medications including terfenadine, quinidine, procainamide, disopyramide, sotalol, bepridil, haloperidol, risperidone, indapamide and flecainide
8. Recent significant hemoptysis (1/2 tea spoon red blood within last month)
9. Concurrent medication that either CYP 450 3A4 inducers or inhibitors
10. Concurrent use of proarrhythmic medications including terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide and flecainide
11. Pregnancy or breast feeding, or patient refusal to use appropriate contraception for female patients in childbirth age
12. Previous malignancy within 5 years, except adequately treated non melanomatous skin cancer or in situ cervical cancer
13. Psychiatric or mental disorder, precluding understanding of the information of the trial related topics and giving valid informed consent
14. Any psychological, familial, geographic or social circumstances which could impair the patient ability to participate in the trial and comply with follow up.
15. Any circumstance which might impair the patient's ability to comply with an out-patient regimen
16. Active uncontrolled infection
17. Serious underlying medical condition (in the judgment of the investigator) which could impair the ability of the patient to participate in the trial
18. Treatment with other experimental drugs within 30 days of entry into the trial
19. Treatment with other anti-cancer therapy
20. Legal incapacity
21. Significant proteinuria (urine protein: creatinine ratio > 1.0)

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2014-12; Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Bevacizumab maximum tolerated dose, in combination with sunitinib | 12 weeks from enrolling patient # 6
  This is the phase I part of the study. patient will enroll on Bevacizumab dose of 5 mg/kg body weight. If no dose limiting toxicity in 1st 6 patients, the dose will be escalated to 10 mg/kg in the remainder of the patients
Assess response rate to the combination of sunitinib and bevacizumab | Through study completion, an average of 6 months
  response rate is the combination of partial response and complete response
Assess the progression free survival on the combination of sunitinib and bevacizumab | up to 5 years
  Progression free survival will be calculated from time of starting therapy till progression or death whichever comes first

SECONDARY OUTCOMES:
Overall survival of patients in this regimen | Participants will be followed for the duration of hospital stay, up to 5 years
  Overall survival will be calculated from date of start on therapy till death
Number of participants with treatment related-adverse effects as assessed by CTCAE v 4.03 | up to 5 years
  toxicity will be graded according to the NCI-CTC version 4.03

CONTACTS AND LOCATIONS:
Overall Officials: Shouki Bazarbashi, MD, Principal Investigator — King Faisal Specialist Hospital & Research Center
Locations (1):
- Oncology Centre, King Faisal Specialist Hospital and Research Centre, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
No- unless the data are so encouraging then this can be done